CLINICAL TRIAL: NCT06771947
Title: Predicting Symptom Trajectories After Thoracoscopic Lung Cancer Surgery Using an Interpretable Machine Learning Model
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Prof., Guangdong Provincial People's Hospital
Other Study IDs: LC-ML
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Machine learning; Patient-reported outcome; Thoracoscopy surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients suffer from a variety of symptoms after thoracoscopic surgery. However, there is a lack of validated predictive tools to identify potentially high-risk patients. This study is anticipated to include approximately 1,500 lung cancer patients who undergo thoracoscopic surgery. Latent class mixed modeling (LCMM) will be used to dentify subgroups of patients with similar symptom trajectories. Machine learning models were developed to predict postoperative symptom trajectories based on collected information. Effective prediction of postoperative symptoms can help identify high-risk patients and take preventive measures.

DETAILED DESCRIPTION:
Thoracoscopic lung cancer surgery is a widely utilized approach for treating early and locally advanced lung cancer. Despite the advantages of thoracoscopic surgery, such as minimal invasion and rapid recovery, patients still suffer from a variety of symptoms such as pain, shortness of breath, sleep disorders or fatigue after surgery, which seriously affects the quality of life. However, there is a lack of validated predictive tools to identify potentially high-risk patients. This study is anticipated to include approximately 1,500 lung cancer patients who undergo thoracoscopic surgery. Patients are invited to fill out the MD Anderson Symptom Inventory-Lung Cancer module after thoracoscopic surgery. Symptoms of interest include pain, shortness of breath, sleep disturbance, and fatigue. Moderate to severe symptoms were defined as a score of ≥ 4. Latent class mixed modeling (LCMM), a clustering technique, can identify subgroups of patients with similar symptom trajectories based on longitudinal patient-reported outcome (PRO) data. Machine learning models were developed to predict postoperative symptom trajectories based on collected information including demographic and clinical information, and operative data. The machine learning models mainly include Random Forest, Support Vector Machines, Neural Networks, XGBoost, etc. The most appropriate model is selected, and model interpretation is performed using the SHAP method. Effective prediction of postoperative symptoms can help identify high-risk patients and take preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old;
* Pathologically diagnosed lung cancer;
* Undergo thoracoscopic surgery, including video-assisted thoracoscopy and robotic-assisted thoracoscopic surgery;
* no prior history of malignancy or lung surgery;
* Have the ability to complete the scale.

Exclusion Criteria:

* Converted to thoracotomy during thoracoscopic surgery;
* Unable to complete the postoperative scale at least two times;
* Missing data values exceeding 30 percent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patient underwent thoracoscopic surgery and completed the MD Anderson Symptom Inventory-Lung Cancer module postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Symptom trajectories after thoracoscopic surgery | Within four weeks after thoracoscopic surgery
  Postoperative symptoms of interest included pain, shortness of breath, sleep disturbances, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, China